CLINICAL TRIAL: NCT06657144
Title: A Phase 1B, Multicenter, Open-Label Study of the Safety and Efficacy of CHS-114 in Combination With Toripalimab With or Without Other Treatments in Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Study of CHS-114 in Combination With Toripalimab and/or Other Treatments in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS-114-102
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Solid Tumor; Advanced Solid Tumor
Keywords: Solid Tumors; Advanced Solid Tumors; Metastatic Solid Tumor; Cancer; Oncology; Tumor; CCR8; PD-1; Gastric cancer; Gastro-esophageal-junction (GEJ) cancer; Esophageal Adenocarcinoma (EAC); Esophageal Squamous Cell Carcinoma; Cisplatin; 5 Fluorouracil (5-FU); Colorectal Carcinoma (CRC)
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Colorectal Neoplasms | interventions — toripalimab; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort A - Arm A1: CHS-114 Dose A + Toripalimab (Experimental): Participants will be treated with dose A of CHS-114 administered as an intravenous (IV) infusion in combination with toripalimab every 3 weeks (Q3W).
  Interventions: Drug: CHS-114; Drug: Toripalimab
- Cohort A - Arm A2: CHS-114 Dose B + Toripalimab (Experimental): Participants will be treated with dose B of CHS-114 administered as an IV infusion in combination with toripalimab Q3W.
  Interventions: Drug: CHS-114; Drug: Toripalimab
- Cohort B - Arm B1: CHS-114 Dose A + Toripalimab (Experimental): Participants will be treated with dose A of CHS-114 administered as an IV infusion in combination with toripalimab Q3W.
  Interventions: Drug: CHS-114; Drug: Toripalimab
- Cohort B - Arm B2: CHS-114 Dose B + Toripalimab (Experimental): Participants will be treated with dose B of CHS-114 administered as an IV infusion in combination with toripalimab Q3W.
  Interventions: Drug: CHS-114; Drug: Toripalimab
- Cohort C - Arm C: CHS-114 Dose B + Toripalimab + 5 fluorouracil (5 FU) + Cisplatin (Experimental): Participants will be treated with dose B of CHS-114 administered as an IV infusion in combination with toripalimab, 5 FU, and cisplatin Q3W.
  Interventions: Drug: CHS-114; Drug: Toripalimab; Drug: 5 Fluorouracil; Drug: Cisplatin
- Experimental: Cohort D - Arm D1 (Liver Mets): CHS-114 + Toripalimab (Experimental): Participants will be treated with CHS-114 administered as an IV infusion in combination with toripalimab Q3W.
  Interventions: Drug: CHS-114; Drug: Toripalimab
- Experimental: Cohort D - Arm D2 (Non-Liver Mets): CHS-114 + Toripalimab (Experimental): Participants will be treated with CHS-114 administered as an IV infusion in combination with toripalimab Q3W.
  Interventions: Drug: CHS-114; Drug: Toripalimab

INTERVENTIONS:
Drug: CHS-114 — Solution for infusion
Drug: Toripalimab — Solution for infusion
Drug: 5 Fluorouracil — Solution for infusion
  Arms: Cohort C - Arm C: CHS-114 Dose B + Toripalimab + 5 fluorouracil (5 FU) + Cisplatin
Drug: Cisplatin — Solution for infusion
  Arms: Cohort C - Arm C: CHS-114 Dose B + Toripalimab + 5 fluorouracil (5 FU) + Cisplatin

SUMMARY:
The main purpose of this study is to evaluate the safety and preliminary efficacy of CHS-114 in combination with toripalimab and/or other standard of care (SOC) compound(s) in participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 1 measurable lesion based on RECIST v1.1 as determined by the Investigator.
* Resolved acute effects of any prior therapy to baseline severity or Grade 1 in accordance with National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5.0, except for adverse events (AEs) not constituting a safety risk per Investigator judgement.

Cohort A (2L Gastric, Gastro-esophageal-junction [GEJ], Esophageal Adenocarcinoma [EAC]) Specific Inclusion Criteria:

* Histologically or cytologically documented unresectable, locally advanced or metastatic gastric, GEJ, or esophageal adenocarcinoma that is human epidermal growth factor receptor 2 (HER2) - negative and microsatellite stable (MSS)/proficient mismatch repair (pMMR).
* Progressed during or after first line systemic therapy that includes a platinum and fluoropyrimidine doublet with or without anti-programmed death receptor 1 (PD-1)/programmed death ligand 1 (PD-L1)-directed therapy (that is, in the second line setting).
* Consent to provide tumor tissue samples (baseline and on-treatment) is required for enrollment.

Cohort B (2L Esophageal Squamous Cell Carcinoma [ESCC]) - Specific Inclusion Criteria:

* Histologically or cytologically documented unresectable, locally advanced or metastatic ESCC.
* Progressed during or after first line systemic therapy including a doublet of platinum and fluoropyrimidine or paclitaxel with or without anti-PD-1/PD-L1-directed therapy or anti-CTLA-4 and anti-PD-1/PD-L1-directed combination therapy.
* Consent to provide results from prior PD-L1 IHC assay score by FDA-approved or equivalent PD-L1 IHC diagnostic tests.
* Consent to provide archival tumor tissue sample (baseline) is required for enrolment.

Cohort C (1L Esophageal Squamous Cell Carcinoma [ESCC]) - Specific Inclusion Criteria:

* Histologically or cytologically documented unresectable, locally advanced or metastatic ESCC.
* Consent to provide baseline tumor tissue is required.
* Consent to provide results from prior PD-L1 IHC assay score by FDA-approved or equivalent PD-L1 IHC diagnostic tests.
* Calculated creatinine clearance ≥60 mL/min.

Cohort D (4L+ Colorectal Carcinoma [CRC]) - Specific Inclusion Criteria:

* Histologically and/or cytologically documented unresectable advanced or metastatic colorectal adenocarcinoma. RAS, BRAF, and microsatellite instability/mismatch repair status for each participant must be documented, according to country level guidelines.
* Participants who have no approved standard therapies with a proven clinical benefit available in the participant's country. These therapies include fluoropyrimidine, oxaliplatin, irinotecan-based chemotherapy, anti-VEGF biological therapy (eg, bevacizumab, aflibercept, ramucirumab), an anti-EGFR therapy (eg, cetuximab, panitumumab) if RAS wildtype unless right-sided, trifluridine/tipiracil or regorafenib, and a BRAF inhibitor (ie, encorafenib) in BRAF V600E mutant).
* Participants who received oxaliplatin in the adjuvant setting and developed metastatic disease during or within 6 months of completing adjuvant therapy are considered eligible without receiving oxalipatin-based therapy in the metastatic setting.
* Consent to provide baseline tumor tissue sample is required for enrolment.

Key Exclusion Criteria:

* History of prior malignancy other than the cancer under study that is progressing or has required active treatment within the past 3 years.
* Symptomatic or untreated central nervous system metastases, including leptomeningeal metastases, requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids.
* Major surgery requiring general anesthesia within 28 days prior to the first dose of study treatment, still recovering from prior surgery, or with surgery scheduled during the study.
* Prior exposure to anti-C-C motif chemokine receptor 8 (CCR8) antibody.
* History of Grade 4 allergic or anaphylactic reaction to any monoclonal antibody (mAb) therapy or any excipient in the study treatment.
* Active uncontrolled bacterial, fungal, or viral infection including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Any condition that, in the opinion of the Investigator or Sponsor, would interfere with the interpretation of study results.

Cohort A (2L Gastric, Gastro-esophageal-junction [GEJ], Esophageal Adenocarcinoma [EAC]) Specific Exclusion Criteria:

* Received ≥ 2 prior systemic anticancer therapies for advanced or metastatic disease.
* Participants at high risk for developing esophageal fistula by clinical assessment or imaging, such as prior history or associated symptoms of esophageal fistula or T4 classification assessed by endoscopic ultrasound (EUS).

Cohort B (2L Esophageal Squamous Cell Carcinoma [ESCC]) - Specific Exclusion Criteria:

* Received ≥ 2 prior systemic anticancer therapies for advanced or metastatic disease.
* Participants at high risk for developing esophageal fistula by clinical assessment or imaging, such as prior history or associated symptoms of esophageal fistula or T4 classification assessed by endoscopic ultrasound (EUS).

Cohort C (1L Esophageal Squamous Cell Carcinoma [ESCC]) - Specific Exclusion Criteria:

* Received ≥ 1 prior systemic anticancer therapies for advanced or metastatic disease.
* Participants who progressed during or within 6 months following the last dose of neoadjuvant, or perioperative therapy with curative intent.
* Participants at high risk for developing esophageal fistula by clinical assessment or imaging, such as prior history or associated symptoms of esophageal fistula or T4 classification assessed by endoscopic ultrasound (EUS).
* Known dihydropyrimidine dehydrogenase deficiency or thymidine synthase gene polymorphism predisposing the participant to 5-FU toxicity.
* Known allergies to 5-FU or cisplatin.

Note: Other protocol-specified inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From first dose of study drug until 90 days after the last dose of study drug (up to approximately 2.25 years)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Based on Investigator Assessment | Up to approximately 2.25 years
  ORR is defined as percentage of participants with confirmed complete response (CR) or partial response (PR) according to RECIST v1.1.
Duration of Response (DOR) Per RECIST v1.1 Based on Investigator Assessment | Up to approximately 2.25 years
  DOR is defined as the time from first documentation of response (CR or PR) to first radiographic documentation of progressive disease or death due to any cause according to RECIST v1.1.
Disease Control Rate (DCR) Per RECIST v1.1 Based on Investigator Assessment | Up to approximately 2.25 years
  DCR is defined as the percentage of participants who achieve a confirmed CR or PR or stable disease (SD) lasting ≥ 12 weeks according to RECIST v1.1.
Progression-free Survival (PFS) Per RECIST v1.1 Based on Investigator Assessment | Up to approximately 2.25 years
  PFS is defined as the time of the first dose of study treatment to the time of the first documented unequivocal disease progression assessed per RECIST v1.1 or death due to any cause (whichever occurs first).
Landmark PFS Rates | Months 6, 9, and 12
Maximum Observed Serum Concentration (Cmax) of CHS-114 | Up to approximately 2.25 years (pre-infusion and up to 336 hours post-infusion)
Time to Reach Cmax (Tmax) of CHS-114 | Up to approximately 2.25 years (pre-infusion and up to 336 hours post-infusion)
Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of CHS-114 | Up to approximately 2.25 years (pre-infusion and up to 336 hours post-infusion)
Number of Participants With Anti-drug Antibodies (ADAs) | Up to approximately 2.25 years

CONTACTS AND LOCATIONS:
Locations (26):
- United States (19):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of Colorado - Aurora Cancer Center, Aurora, Colorado
  - Winship Cancer Center - Emory University, Atlanta, Georgia
  - Ochsner Health, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Christus St Vincent Regional Medical Center, Santa Fe, New Mexico
  - START New York, Lake Success, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburg Medical Center _UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Central South, Austin, Texas
  - START San Antonio, LLC., San Antonio, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - START Mountain Region, LLC., West Valley City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Taiwan (7):
  - E-Da Cancer Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Kapoor VN, Chin DJ, Klakamp SL, Baruffaldi F, Mohan JF, Haines R, Dulak A, Panduro M, Ren Y, Masia R, Hill JA, LaVallee TM, Rajasekaran N. CHS-114: an afucosylated anti-CCR8 monoclonal antibody that selectively depletes intratumoral Treg cells and induces antitumor immune responses. Mol Cancer Ther. 2025 Dec 22. doi: 10.1158/1535-7163.MCT-25-0367. Online ahead of print. PMID 41423415